CLINICAL TRIAL: NCT05222451
Title: Nutritional Strategies to Enhance Lung Function in Asthmatics with Obesity
Brief Title: Nutrition for Asthmatics with Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Jacob T. Mey, PhD RD, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: PBRC 2022-001 A
Record Dates: First submitted 2022-01-05; First posted 2022-02-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Asthma; Obesity
Keywords: ketone; diet; metabolism
MeSH Terms: conditions — Asthma; Obesity; Ketosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be made aware of the diet allocation. However, due inherent differences in macronutrient content of the diets, participants may perceive differences in the quantity of various food groups or in the taste, texture or smell of foods present in the diet. To address this, diets will be designed to minimize noticeable differences for the participant. The investigator and outcomes assessor will remain fully masked to diet provision.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dietary Guidelines for Americans (Experimental): 7 days of a diet consistent with the Dietary Guidelines for Americans (DGA).
  Interventions: Other: DGA Diet
- Medium Chain Triglyceride Supplemented DGA (Experimental): 7 days of a diet consistent with the Dietary Guidelines for Americans supplemented with medium chain triglycerides (MCT).
  Interventions: Other: MCT Diet
- Ketogenic Diet (Experimental): 7 days of a ketogenic diet (KETO).
  Interventions: Other: KETO Diet

INTERVENTIONS:
Other: DGA Diet — A fully provisioned isocaloric, isonitrogenous study diet following the Dietary Guidelines for Americans (DGA)
  Including:
  * A variety of vegetables and fruits
  * Grains, at least half of which are whole grains
  * Fat-free or low-fat dairy
  * A variety of protein foods, including seafood, lean meats and poultry, eggs, legumes, nuts, and seeds
  * This healthy eating pattern also limits saturated fats and trans fats, added sugars, and sodium.
  Arms: Dietary Guidelines for Americans
Other: MCT Diet — A fully provisioned isocaloric, isonitrogenous study diet following the Dietary Guidelines for Americans supplemented with medium chain triglycerides (MCT).
  Arms: Medium Chain Triglyceride Supplemented DGA
Other: KETO Diet — A fully provisioned isocaloric, isonitrogenous ketogenic study diet.
  Arms: Ketogenic Diet

SUMMARY:
This study will test the effect of diet on asthma in individuals with obesity.

DETAILED DESCRIPTION:
This is a crossover design pilot trial that will recruit 12 adults with obesity and asthma. Participants will undergo screening and a lead-in period before being randomized to a series of three, 7-day diets with a 7+ day washout period between each diet. Asthma control and lung function will be assessed at the completion of each diet.

The goal of this pilot trial is to understand the effect of diet on asthma and conduct an exploratory analysis on factors that may predict the response to diet.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* BMI: 30-45 kg/m2
* asthma diagnosed by medical specialist (confirmed in medical history)
* partly controlled or uncontrolled asthma by Asthma Control Test score ≤22
* owns a device compatible with ZEPHYRx platform
* stable asthma medication use (no change in the past 2 months).

Exclusion Criteria:

* Diabetes or using diabetes medications that may lower blood glucose levels
* point of care fasting blood glucose ≥126 mg/dl or triglycerides ≥400 mg/dl
* current smoking or smoking history of greater than 10 pack-years
* other significant respiratory or cardiac disease or the presence of clinically important comorbidities, e.g., COPD, renal failure, liver disease; uncontrolled hypertension defined as systolic blood pressure ≥160 mm/Hg, or diastolic blood pressure ≥100 mm/Hg
* pregnant or nursing women
* food preferences or allergies inconsistent with study diet capabilities
* noncompliance with lead-in period requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Asthma Control | Baseline
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.
Asthma Control | After 7 days on Diet#1
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.
Asthma Control | After 7 days on Diet#2
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.
Asthma Control | After 7 days on Diet#3
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.

SECONDARY OUTCOMES:
Lung Function | Baseline
  FEV1 (forced expiratory volume in 1 second; % of predicted)
Lung Function | After 7 days on Diet#1
  FEV1 (forced expiratory volume in 1 second; % of predicted)
Lung Function | After 7 days on Diet#2
  FEV1 (forced expiratory volume in 1 second; % of predicted)
Lung Function | After 7 days on Diet#3
  FEV1 (forced expiratory volume in 1 second; % of predicted)
FENO | Baseline
  FENO (ppm)
FENO | After 7 days on Diet#1
  FENO (ppm)
FENO | After 7 days on Diet#2
  FENO (ppm)
FENO | After 7 days on Diet#3
  FENO (ppm)
FEV1/FVC | Baseline
  FEV1/Forced Vital Capacity (FVC) ratio
FEV1/FVC | After 7 days on Diet#1
  FEV1/Forced Vital Capacity (FVC) ratio
FEV1/FVC | After 7 days on Diet#2
  FEV1/Forced Vital Capacity (FVC) ratio
FEV1/FVC | After 7 days on Diet#3
  FEV1/Forced Vital Capacity (FVC) ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Mey, PhD, RD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Study data will be provided upon request and approval by study PI.